CLINICAL TRIAL: NCT00740272
Title: Af Ablation In Brady-Tachy Syndrome
Acronym: Alternative
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJM-FR01
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Brady-tachy Syndrome
Keywords: brady-tachy syndrome; AF ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AF ablation + pacemaker
  Interventions: Procedure: AF ablation + pacemaker implantation
- 2 (Active Comparator): Pacemaker
  Interventions: Procedure: Pacemaker implantation

INTERVENTIONS:
Procedure: AF ablation + pacemaker implantation — regular pacemaker implantation and concomitant AF ablation procedure (PV isolation)
  Arms: 1
Procedure: Pacemaker implantation — regular pacemaker implantation
  Arms: 2

SUMMARY:
The aim of the study is to evaluate the impact of atrial fibrillation ablation in patients presenting a brady-tachy syndrome on the AF burden.

The hypothesis of the study is that AF ablation prevents not only from AF episodes recurrence but also from bradycardic episodes.

DETAILED DESCRIPTION:
The study is a randomized study 1:1 AF ablation vs non AF ablation. Patients are followed for 1 year. 38 patients will be required to show a significant reduction in AF burden.

ELIGIBILITY:
Inclusion Criteria:

* paroxystic AF
* symptomatic pauses (>5s at night or 3s during daytime)

Exclusion Criteria:

* permanent AF
* age > 80 y
* pregnant women
* minors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
AF burden | 1 year

SECONDARY OUTCOMES:
Quality of life | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital St joseph, Marseille
  - CHU, Rouen
  - Clinique Pasteur, Toulouse